CLINICAL TRIAL: NCT05826353
Title: A Double-Masked, Randomized, Placebo-Controlled, Parallel-Group, 12-Week Administration With Two-Week Gradual Dose Taper Phase and 38-Week Follow-Up Phase, Phase 3 Study to Investigate the Safety and Efficacy of Ripasudil (K-321) Eye Drops After Simultaneous Cataract Surgery and Descemetorhexis in Subjects With Fuchs Endothelial Corneal Dystrophy
Brief Title: A Study to Investigate the Safety and Efficacy of K-321 Eye Drops After Simultaneous Cataract Surgery and Descemetorhexis in Participants With Fuchs Endothelial Corneal Dystrophy (FECD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-321-303
Record Dates: First submitted 2023-04-06; First posted 2023-04-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Fuchs Endothelial Corneal Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy | interventions — K-115

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- K-321 (Experimental): K-321 ophthalmic solution four times daily (QID) for 12 weeks followed by a two-week gradual dose taper phase and 38-week follow-up phase
  Interventions: Drug: Ripasudil
- Placebo (Placebo Comparator): Placebo ophthalmic solution QID for 12 weeks followed by a two-week gradual dose taper phase and 38-week follow-up phase
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ripasudil — K-321 ophthalmic solution
  Other Names: K-321
  Arms: K-321
Drug: Placebo — Placebo ophthalmic solution
  Arms: Placebo

SUMMARY:
A study to assess the safety and efficacy of K-321 in participants with FECD after simultaneous cataract surgery and descemetorhexis.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years old at the screening visit (Visit 1)
* Has a diagnosis of FECD at Visit 1
* Meet all other inclusion criteria outlined in the Clinical Study Protocol.

Exclusion Criteria:

* Is a female subject of childbearing potential and any of the following is true:

  1. is pregnant or lactating/breastfeeding, or
  2. is not surgically sterile, not post-menopausal (no menses for the previous 12 months), or not practicing an effective method of birth control as determined by the Investigator (eg, oral contraceptives, double barrier methods, hormonal injectable or implanted contraceptives, tubal ligation, or partner with vasectomy)
* Meet any other exclusion criteria outlined in the Clinical Study Protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Time to improvement in best corrected (distance) visual acuity (BCVA) by ETDRS letter score during the first 12 weeks | Baseline to Week 12

SECONDARY OUTCOMES:
Time to improvement in best corrected (distance) visual acuity (BCVA) by ETDRS letter score during the first 12 weeks | Baseline to Week 12
Time to achievement in best corrected (distance) visual acuity (BCVA) by ETDRS letter score during the first 12 weeks | Baseline to Week 12
Central corneal Endothelial Cell Density (ECD) (cells/mm2) at Week 12 | Week 12
  Central corneal endothelial cell images will be captured by non-contact specular microscopy.
Time to achievement of no corneal edema during the first 12 weeks | Baseline to Week 12
Time to exceed in BCVA pre-DSO ETDRS letter score during the first 12 weeks | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Shona Pendse, MD, MMSc, Study Chair — Kowa Pharma Development Co.
Locations (43):
- United States (21):
  - Keck Hospital of USC, Los Angeles, California
  - Macy Eye Center, Los Angeles, California
  - Byers Eye Institute at Stanford, Palo Alto, California
  - Sacramento Eye Consultants, Sacramento, California
  - Gorovoy MD Eye Specialists, Fort Myers, Florida
  - Bascom Palmer Eye Institute, Palm Beach Gardens, Florida
  - Grene Vision Group-Wichita, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - W Kellogg Eye Center, Ann Arbor, Michigan
  - Verdier Eye Center, Grand Rapids, Michigan
  - Vance Thompson Vision - Omaha, Omaha, Nebraska
  - Eye Associates of New Mexico - Albuquerque - Northside, Albuquerque, New Mexico
  - NYU Langone Health, New York, New York
  - Vance Thompson Vision West Fargo, West Fargo, North Dakota
  - Cincinnati Eye Institute-1945 Cei Dr, Blue Ash, Ohio
  - University Hospitals Cleveland Medical Center - 11100 Euclid Ave, Cleveland, Ohio
  - Devers Eye Institute, Portland, Oregon
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Eye Associates, Houston, Texas
  - R and R Eye Research, LLC., San Antonio, Texas
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- Canada (3):
  - Dr. Greg Moloney, Vancouver, British Columbia
  - Prism Eye Institute - Mississauga-Oakville, Oakville, Ontario
  - Precision Cornea Centre, Ottawa, Ontario
- Denmark (2):
  - Rigshospitalet Glostrup-Valdemar Hansens Vej 1-23, Glostrup Municipality, Capital
  - Aarhus Universitetshospital, Aarhus N, Central Jutland
- Germany (7):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitatsklinkum Erlangen-Ulmenweg 18, Erlangen, Bavaria
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - Universitatsklinikum Dusseldorf, Düsseldorf, North Rhine-Westphalia
  - Universität des Saarlandes, Homburg, Saarland
  - LMU Klinikum der Universität, München
- Spain (7):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Althaia Xarxa Assistencial Universitaria Manresa, Manresa, Barcelona
  - Hospital Arruzafa, Córdoba, Córdoba
  - Instituto Oftalmologico Fernandez Vega, Oviedo, Principality of Asturias
  - Oftalvist - Barcelona, Barcelona
  - Institut Catala de Retina (ICR), Barcelona
  - Instituto de Microcirugia Ocular, Barcelona
- United Kingdom (3):
  - The Royal Liverpool University Hospital, Liverpool, Lancashire
  - Moorfields Eye Hospital, London, London, City of
  - Royal Victoria Infirmary, Newcastle upon Tyne, Tyne and Wear